CLINICAL TRIAL: NCT03595345
Title: A Worldwide Usable Scoring System for Patients With Hepatocellular Cancer Waiting for Liver Transplantation
Brief Title: A Worldwide Score for Hepatocellular Cancer and Liver Transplantation
Acronym: TRAIN-SCORE
Status: Completed | Type: Observational
Sponsor: European Hepatocellular Cancer Liver Transplant Group (Other)
Responsible Party: Principal Investigator, Quirino Lai, Principal investigator and Data manager of the EurHeCaLT Study Group, European Hepatocellular Cancer Liver Transplant Group
Other Study IDs: #0001
Record Dates: First submitted 2018-07-11; First posted 2018-07-23 (Actual); Last update posted 2018-10-29 (Actual); Status verified 2018-10

CONDITIONS: Liver Cancer; Dropout, Patient; Recurrence
Keywords: delisting; tumor-specific death; Milan Criteria
MeSH Terms: conditions — Liver Neoplasms; Patient Dropouts; Recurrence | interventions — Liver Transplantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Training set: 2200 HCC cases from East and West centres enlisted for LT and then delisted or transplanted
  Interventions: Procedure: Liver transplantation
- West validation set: 630 HCC cases from a Western centre enlisted for LT and then delisted or transplanted
  Interventions: Procedure: Liver transplantation
- East validation set: 300 HCC cases from a Eastern centre enlisted for LT and then delisted or transplanted
  Interventions: Procedure: Liver transplantation

INTERVENTIONS:
Procedure: Liver transplantation — Liver transplantation

SUMMARY:
The present study has been developed with multiple aims: 1) to refine available models for liver transplantation which would be able to cover the fate of HCC candidates from an ITT point of view; 2) to develop such an approach on cohorts coming from both Eastern and Western countries; 3) to maintain simplicity of use; 4) to provide individual prognostication taking into account different causes of death, through a competing-risk model; 5) to provide an external validation on cohorts coming from both Eastern and Western countries. All these aims converge at providing a comprehensive and useful assessment suitable for both candidates selection and allocation priority.

DETAILED DESCRIPTION:
For two decades, the Milan Criteria (MC) have represented the cornerstone in the selection of patients with hepatocellular cancer (HCC) as candidates for liver transplantation (LT). Since then, several Western and Eastern centres have tried to overcome MC stringency with the aim to expand the number of potentially transplantable patients without increasing the risk of post-LT tumour recurrence. Recently, variables correlated with HCC biology have been introduced to capture its aggressiveness and suitability for LT. Among the most commonly proposed, we can cite the alpha-fetoprotein (AFP) and the radiological response after neo-adjuvant loco-regional treatments (LRT). The effort to combine HCC morphology and biology is now emerging as the more promising approach for further refining the selection process of HCC candidates. The recently proposed prognostic indexes Metroticket 2.0, Time-Radiological-response-Alpha-fetoprotein-INflammation (TRAIN), Model Of Recurrence After Liver transplant (MORAL) and French AFP-model represent the most promising results of such planned endeavours.

With the intent to be clinically useful, a prognostic system must achieve not only the most common performance metrics, such as discrimination and calibration, but also an adequate coverage of the population in which it would be applied. It can be argued that a prognostic system based only on criteria available at the moment of LT could not satisfy such a pre-requisite when the entire population of HCC patients waiting in the list for LT is taken into account, considering an intention-to-treat (ITT) point of view. In this sense, only the TRAIN system developed an ITT analysis, whereas the remaining were all based on pre-transplant information. The second quality that a clinically useful prognostic system should have is its immediacy. Thus, it should be based on commonly available information, not requiring additional analyses or exams if not justified by a substantial improvement in accuracy. Last but not least, a prognostic system should also provide for an individual prediction in addition to risk-stratification, with the intent to offer personalized prognostication for each different patient. To date, only the Metroticket 2.0 fulfils these two last requisites. A final important quality of the Metroticket 2.0 is that it applied a competing-risk analysis able to clean up the HCC-related cause of death from other non-tumour-related causes.

On this background, we developed the present study with multiple aims: 1) to refine available models which would be able to cover the fate of HCC candidates from an ITT point of view; 2) to develop such an approach on cohorts coming from both Eastern and Western countries; 3) to maintain simplicity of use; 4) to provide individual prognostication taking into account different causes of death, through a competing-risk model; 5) to provide an external validation on cohorts coming from both Eastern and Western countries. All these aims converge at providing a comprehensive and useful assessment suitable for both candidates selection and allocation priority.

ELIGIBILITY:
Inclusion Criteria:

* All the adult ((≥18 years) patients enlisted for liver transplant with the radiological/histological diagnosis of hepatocellular cancer during the period 01/01/2000-31/03/2017

Exclusion Criteria:

* Mixed hepatocellular-cholangiocellular
* Cholangiocellular cancer misdiagnosed as HCC
* Post-LT incidental HCC.
* Patients enlisted before 01/01/2000

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The participating centers for the creation of the training set cohort were: Brussels (Belgium; n=355), New York Columbia University/Weill Cornell Medical Center (USA; n=353), Innsbruck (Austria; n=330), New Delhi (India; n=270), Rome Sapienza University (Italy; n=265), Kyoto (Japan; n=230), Taiwan (Republic of China; n=200), Mainz (Germany; n=176), Kyushu (Japan; n=161), and Hangzhou Shulan Health Hospital/First Affiliated Hospital (Popular Republic of China; n=94).
  For the testing/external cohort, two additional centres participated to the study, namely the Western center from Padua (Italy; n=630) and the Easter center from Hong Kong (n=330) applying the same inclusion/exclusion criteria as for the training cohort.
Sampling Method: Non-Probability Sample
Enrollment: 3100 (Actual)
Dates: Start 2016-12-15 (Actual); Primary Completion 2018-10-15 (Actual); Study Completion 2018-10-15 (Actual)

PRIMARY OUTCOMES:
Tumour-specific death | 5 years after transplant
  Death for recurrence or other HCC-related causes

SECONDARY OUTCOMES:
Drop-out | 1 year after waiting list inscription
  Drop-out for death or HCC progression

CONTACTS AND LOCATIONS:
Locations (1):
- UCL, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: Undecided